CLINICAL TRIAL: NCT04198896
Title: Clinical Aspects of Atherosclerotic-Carcinogenesis Hypothesis
Brief Title: The Sakakibara Health Integrative Profile of Atherosclerotic-Carcinogenesis Hypothesis (SHIP-AC)
Acronym: SHIP-AC
Status: Completed | Type: Observational
Sponsor: Sakakibara Heart Institute (Other)
Responsible Party: Principal Investigator, Makoto Suzuki, Director, Department of Cardiology, Sakakibara Heart Institute
Other Study IDs: SHIP03
Record Dates: First submitted 2019-12-08; First posted 2019-12-13 (Actual); Last update posted 2019-12-18 (Actual); Status verified 2019-12

CONDITIONS: Cancers; Atheroscleroses, Coronary; Atherosclerosis of Artery
Keywords: Atherosclerosis, cancers
MeSH Terms: conditions — Neoplasms; Coronary Artery Disease; Atherosclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1095 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CAD-only: patients with diagnosed coronary artery diseases (CAD) without any other atherosclerotic cardiovascuar diseases at the entry of SHIP
  Interventions: Other: incidece of cancers
- CAD with poly-arterial diseases: patients with diagnosed coronary artery diseases (CAD) with other atherosclerotic cardiovascuar diseases such as any of aortic and/or peripheral artery diseases at the entry of SHIP
  Interventions: Other: incidece of cancers

INTERVENTIONS:
Other: incidece of cancers — With a continuous surveillance system to track all subsequent incidents of cardiovascular diseases and/or non-cardiovascular diseases via direct contact in the outpatient department, hospital records, and a mailed questionnaire at least once a year, an incidence of cancers was identified

SUMMARY:
As previously reported (IJC Heart & Vasculature 2017; 17: 11.), our epidemiological analysis showing high incidence of cancers in patients with atherosclerotic cardiovascular diseases as compared with those with non-atherosclerotic cardiovascular diseases may imply a clinical possibility of a role of atherosclerosis in cancer developments. In the present study, to address our hypothesis that cancer developments may come with a strength of atherosclerosis, we traced an incidence of cancers in a total of 8,856 patients with coronary artery diseases (CAD) for a median follow-up of 1,095 days (interquartile range, 719-1,469 days) using the Sakakibara Health Integrative Profile (SHIP) database.

DETAILED DESCRIPTION:
In accordance with a presence or absence of poly-arterial diseases such as aortic and/or peripheral artery diseases as an indicator of a strength of atherosclerosis, an incidence of cancers and all-cause death in two cohorts of 8,140 patients with CAD-only and 716 with CAD with poly-arterial diseases were evaluated to track an incidence of cancers and ali-cause mortality during median follou-up periods of 3 to 4 years.

ELIGIBILITY:
Inclusion Criteria:

* patients with diagnosed coronary artery diseases without a dignosis of cancers at the entry of SHIP between January 2009 and July 2014.

Exclusion Criteria:

* patients with diagnosed coronary artery diseases who had already been diagnosed with any cancers at the time of enrollment in the SHIP, and who were not followed-up after the entry of SHIP.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: same as eligibility criteria
Sampling Method: Non-Probability Sample
Enrollment: 8856 (Actual)
Dates: Start 2009-01 (Actual); Primary Completion 2019-10 (Actual); Study Completion 2019-10 (Actual)

PRIMARY OUTCOMES:
inicidence of cancers | through study completion, an average of 3 years
  number of all types of cancers during follow-up periods

SECONDARY OUTCOMES:
all-cause mortality | through study completion, an average of 3 years
  number of all types of death during follow-up periods

IPD SHARING:
Plan to Share IPD: No
After completed, the data will be shared with simlar study investigators over the world

REFERENCES:
- [Derived] Suzuki M, Tomoike H, Dai Z, Hosoda T, Sumiyoshi T, Hosoda S, Isobe M. Polyvascular Disease and the Incidence of Cancer in Patients with Coronary Artery Disease. JMA J. 2022 Oct 17;5(4):498-509. doi: 10.31662/jmaj.2022-0098. Epub 2022 Sep 26. PMID 36407071